CLINICAL TRIAL: NCT03457012
Title: SURE CANADA: A Multi-centre, Prospective, Noninterventional Study Investigating the Effectiveness of Once Weekly Subcutaneous Semaglutide in a Real World Adult Population With Type 2 Diabetes
Brief Title: A Research Study Looking at How Semaglutide Works in People With Type 2 Diabetes in Canada, as Part of Local Clinical Practice
Acronym: SURE CANADA
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9535-4428; U1111-1205-5853 (Other: World Health Organisation (WHO))
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Semaglutide: Participants will receive semaglutide at the treating physician's discretion as part of the usual clinical practice. The prescription and use of semaglutide is completely independent of this study. Total study duration for the individual patient will be approximately 30 weeks
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Patients will be treated with commercially available semaglutide in a prefilled pen injector (FlexTouch® variant) according to routine local clinical practice at the discretion of the treating physician. Other anti-hyperglycaemic treatments will be prescribed at the physician's discretion.

SUMMARY:
The purpose of the study is to collect information on how semaglutide works in real world patients. Participants will get semaglutide prescribed by the study doctor. The study will last for about 6 to 8 months. Participants will be asked to complete some questionnaires about the health and the diabetes treatment. Participants will complete these during the normally scheduled visits with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study-related activities (study-related activities are any procedures related to recording of data according to protocol)
* The decision to initiate treatment with commercially available semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study
* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Diagnosed with type 2 diabetes at least 12 weeks prior to inclusion
* Available and documented HbA1c value less than or equal to 12 weeks prior to initiation of semaglutide treatment

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Treatment with any investigational drug within 90 days prior to enrolment into the study
* Hypersensitivity to semaglutide or to any of the excipients

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with type 2 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Change in Glycated Haemoglobin A1c (HbA1c) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28-38)
  Measured in % points
Change in HbA1c | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28-38)
  Measured in mmol/mol

SECONDARY OUTCOMES:
Change in body weight | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28-38)
  Measured in kg
Change in body weight | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28-38)
  Measured in %
Change in waist circumference | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28-38)
  Measured in cm
HbA1c level at end of study: < 8.0% (64 mmol/mol) (yes/no) | At end of study (week 28-38)
  Number of participants who achieved/not achieved HbA1c level at end of study: <8.0%
HbA1c level at end of study: <7.5% (59 mmol/mol) (yes/no) | At end of study (week 28-38)
  Number of participants who achieved/not achieved HbA1c level at end of study: <7.5%
HbA1c level at end of study: <7.0% (53 mmol/mol) (yes/no) | At end of study (week 28-38)
  Number of participants who achieved/not achieved HbA1c level at end of study: <7.0%
Reduction in HbA1c of 1.0% point or more (yes/no) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28-38)
  Number of participants who achieved/not achieved reduction in HbA1c of 1.0% point or more
Weight reduction of 3.0% or more (yes/no) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28-38)
  Number of participants who achieved/not achieved weight reduction of 3.0% or more
Weight reduction of 5.0% or more (yes/no) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28-38)
  Number of participants who achieved/not achieved weight reduction of 5.0% or more
HbA1c reduction of 1.0% point or more and weight reduction of 3.0% or more (yes/no) | Baseline (up to 12 weeks prior to treatment initiation at week 0), end of study (week 28-38)
  Number of participants who achieved/not achieved HbA1c reduction of 1.0% point or more and weight reduction of 3.0% or more
Patient reported severe or documented hypoglycaemia (yes/no) | Between baseline (week 0) and end of study (week 28-38)
  Number of participants who reported/not reported severe or documented hypogycaemia
Change in Diabetes Treatment Satisfaction Questionnaire - Status (DTSQs) (absolute treatment satisfaction): Total treatment satisfaction | Baseline (week 0), end of study (week 28-38)
  The status version (DTSQs) provides a measure of how satisfied patients are with their current diabetes treatment. It consists of 8 questions, which are to be answered on a Likert scale from 0 to 6 (0 = very dissatisfied to 6 = very satisfied). Six questions are summed to produce a total Treatment Satisfaction score. The remaining two questions are concerning perceived frequency of hyperglycaemia and perceived frequency of hypoglycaemia, respectively.
Change in Diabetes Treatment Satisfaction Questionnaire - Change (DTSQc) (relative treatment satisfaction): Total treatment satisfaction | Baseline (week 0), end of study (week 28-38)
  The change version (DTSQc) has the same 8 items as the status version, but is reworded to direct the patients to compare the experience of the current treatment with the experience of previous treatment. Each question is scored on a scale of -3 to +3 (-3 = much less satisfied now to +3 = much more satisfied now), with 0 (midpoint), representing no change.
Change in Short Form (SF)-36 v2: Physical summary component | Baseline (week 0), end of study (week 28-38)
  The SF-36®v2 questionnaire has 36 questions grouped into eight domains termed: physical functioning, bodily pain, role-physical, general health, vitality, social functioning, role-emotional and mental health, which again can be combined to give two summary component scores (overall mental- and physical health).
Change in SF-36 v2: Mental summary component | Baseline (week 0), end of study (week 28-38)
  The SF-36®v2 questionnaire has 36 questions grouped into eight domains termed: physical functioning, bodily pain, role-physical, general health, vitality, social functioning, role-emotional and mental health, which again can be combined to give two summary component scores (overall mental- and physical health).
Patient completed the study under treatment with semaglutide (yes/no) | At end of study (week 28-38)
  Number of patients who completed/not completed the study under treatment with semaglutide

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Cambridge, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://www.novonordisk-trials.com

REFERENCES:
- [Result] Yale JF, Catarig AM, Grau K, Harris S, Klimek-Abercrombie A, Rabasa-Lhoret R, Reardon L, Woo V, Liutkus J. Use of once-weekly semaglutide in patients with type 2 diabetes in routine clinical practice: Results from the SURE Canada multicentre, prospective, observational study. Diabetes Obes Metab. 2021 Oct;23(10):2269-2278. doi: 10.1111/dom.14468. Epub 2021 Aug 15. PMID 34142429
- [Derived] Yale JF, Bodholdt U, Catarig AM, Catrina S, Clark A, Ekberg NR, Erhan U, Holmes P, Knudsen ST, Liutkus J, Sathyapalan T, Schultes B, Rudofsky G. Real-world use of once-weekly semaglutide in patients with type 2 diabetes: pooled analysis of data from four SURE studies by baseline characteristic subgroups. BMJ Open Diabetes Res Care. 2022 Apr;10(2):e002619. doi: 10.1136/bmjdrc-2021-002619. PMID 35383100